CLINICAL TRIAL: NCT06609954
Title: "COMPARATIVE EFFECTS of REDUCED EXERTION HIGH INTENSITY TRAINING (REHIT) VERSUS HIGH INTENSITY INTERVAL TRAINING (HIIT) on ANTHROPOMETRIC MEASURES in OVERWEIGHT and OBESE ADULTS"
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/26
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-08

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial having two groups. One group(interventional group) will be given Reduced Exertion High Intensity Training (REHIT) and the other group (control group) will be given High intensity Interval Training (HIIT).
Who Masked: Participant
Masking Description: single-blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reduced Exertion High intensity Training (REHIT) Group (Experimental): Participant will perform a 5 min warm-up exercises then do cycling or treadmill running for 20 min at 40%-60% of HRR and then will conclude with 5 min cool down exercises. From week 2 to 6 participants will be instructed to perform training sessions on a cycle ergometer.A 3-minute cool-down period will conclude each session. Patients in this group will be provided with a caloric restriction plan by a nutritionist that will be followed throughout the training duration.
  Interventions: Other: Reduced Exertion High Intensity Training (REHIT)
- High Intensity Interval Training (HIIT) (Experimental): Participant will perform a 5 min warm-up exercises then do cycling or treadmill running for 20 min at 40%-60% of HRR and then will conclude with 5 min cool down exercises. From week 2 to 6 participants will be instructed to perform a warm up of 5 min, then 4 bouts of 4 min of HIIT will be performed at 80%-95% of HRR separated by 3-min active recovery periods of moderate intensity cycling at 60%-70% of the HRR followed by 5 min cool down exercises. Patients in this group will be provided with a caloric restriction plan by a nutritionist that will be followed throughout the training duration.
  Interventions: Other: High Intensity Interval Training (HIIT)

INTERVENTIONS:
Other: Reduced Exertion High Intensity Training (REHIT) — Participant will perform a 5 min warm-up exercises then do cycling or treadmill running for 20 min at 40%-60% of HRR and then will conclude with 5 min cool down exercises. From week 2 to 6 participants will be instructed to perform training sessions on a cycle ergometer. Each session will consist of a 3-minute warm-up period followed by two 20-second all-out sprints interspersed with 3 minutes of slow pedaling for recovery. Total of 18 sessions of REHIT will be performed thrice a week on alternate days by the participants for consecutive 6 weeks.
  Arms: Reduced Exertion High intensity Training (REHIT) Group
Other: High Intensity Interval Training (HIIT) — Patients in this group will be provided with a caloric restriction plan by a nutritionist that will be followed throughout the training duration. Week 1 will be baseline fitness level and familiarization week. Participant will perform a 5 min warm-up exercises then do cycling or treadmill running for 20 min at 40%-60% of HRR and then will conclude with 5 min cool down exercises. From week 2 to 6 participants will be instructed to perform a warm up of 5 min, then 4 bouts of 4 min of HIIT will be performed at 80%-95% of HRR separated by 3-min active recovery periods of moderate intensity cycling at 60%-70% of the HRR followed by 5 min cool down exercises. Pre and post session vitals will be noted. Total of 18 sessions of either HIIT will be performed thrice a week on alternate days by the participants for consecutive 6 weeks.
  Arms: High Intensity Interval Training (HIIT)

SUMMARY:
Obesity is a global health concern associated with an increased risk of cardio-metabolic diseases and reduced overall health. Exercise is a proven modality for managing obesity, with current focus of researches on identifying more time-efficient modes of exercise training. REHIT and HIIT have proven benefits but comparative effects of REHIT and HIIT in overweight and obese adults is yet to be determined. Hence the objective of this study is to compare the effects of reduced exertion high intensity training (REHIT) versus high intensity interval training (HIIT) on anthropometric measures (weight, waist circumference, hip circumference, waist-to-hip ratio), CUN-BAE adiposity index and cardiorespiratory fitness in overweight and obese adults.

DETAILED DESCRIPTION:
Obesity is a global health concern associated with an increased risk of cardio-metabolic diseases and reduced overall health. Exercise is a proven modality for managing obesity, with current focus of researches on identifying more time-efficient modes of exercise training. REHIT and HIIT have proven benefits but comparative effects of REHIT and HIIT in overweight and obese adults is yet to be determined.The significance of this study is to compare the effects of reduced exertion high intensity training (REHIT) versus high intensity interval training (HIIT) and will also investigate the effectiveness of REHIT as an alternative for overweight and obese individuals who perceive HIIT as too demanding. If found effective, it can also help in providing training protocol for optimizing cardiovascular health in this population, potentially leading to improved outcomes and reduced healthcare burdens. The results of this study will also add data to literature regarding the effects of REHIT and HIIT on anthropometric measures in overweight and obese. Main objective of this study is to compare the effects of reduced exertion high intensity training (REHIT) versus HIIT on anthropometric measures (weight, waist circumference, hip circumference, waist-to-hip ratio), CUN-BAE adiposity index and Cardiorespiratory fitness in overweight and obese individuals. The participants meeting the eligibility criteria will be recruited followed by random allocation to one of the 2 groups, following which they will be required to complete a self-reported demographic form and will be screened using Physical Activity Readiness Questionnaire (PAR-Q). Baseline evaluation will be done using tape measure for anthropometric, assessment of waist circumference and hip circumference, CUN-BAE index for adiposity and Queen's College step test for cardio-respiratory fitness. Experimental group A will perform REHIT while experimental group B will perform HIIT. Participants will also be provided with dietary restriction plan that will be followed during the training protocol. Exercise training would be performed for consecutive 6 weeks, 3 times a week on alternative days for total of 18 sessions.

ELIGIBILITY:
Inclusion Criteria

* Both male and female adults aged 18-45 years
* Overweight individuals with BMI ≥ 23kg/m²- 24.9kg/m²
* Obese individuals with BMI ≥ 25kg/m²
* Individuals falling in low PA category as per IPAQ Exclusion Criteria
* Individuals with any diagnosed cardiovascular, metabolic or pulmonary disease
* Current neurological or musculoskeletal conditions which limit participation in the study
* Any active infections
* Those with any contraindication to exercise testing or training.
* Currently following any dietary restriction plans for weight loss

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Waist circumference | 6 weeks
  Will be measured using a cloth tape measure. Waist circumference will be measured at the level of the smallest circumference above the umbilicus and below the xiphoid appendix.
Hip Circumference: | 6 weeks
  Measure at the widest point of the hips, with feet together
Waist-to-hip Ratio: | 6 weeks
  To determine the waist-to-hip ratio, divide the WC by the HC
Cardiorespiratory fitness | 6 weeks
  Cardiorespiratory Fitness will be assessed via Queens College step test.
Adiposity index | 6 weeks
  Evaluation will be done using CUN-BAE INDEX (Clínica Universidad de Navarra-Body Adiposity Estimator)

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan